CLINICAL TRIAL: NCT03939169
Title: The Efficiency of Using Supportive Postures and Holding Techniques in Order to Minimize Premature Infant Pain During Naso-gastric Tube Insertion, in the Presence or Absence of the Mother.
Brief Title: The Efficiency of Using Supportive Postures and Holding Techniques to Minimize Premature Infant Pain (PAP)
Acronym: PAPS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in Principal Investigator Role
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-07-CHRMT
Record Dates: First submitted 2019-04-30; First posted 2019-05-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Premature Infant
Keywords: pain; naso-gastric tube
MeSH Terms: conditions — Premature Birth; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Skin-to-skin support (Other): The newborn is dressed in one layer of clothing with a hat, he is placed in the ventral position directly on the mother's chest, covered with a warm blanket and held in place with a band during the insertion of the naso-gastric feeding tube.
  Interventions: Other: Installation of a naso-gastric feeding tube
- Holding (Other): The newborn is held in his mother's arms during insertion of the naso-gastric feeding tube.
  Interventions: Other: Installation of a naso-gastric feeding tube
- Four hands care (Other): Carried out by two professionals: one health-care professional supports the child and helps stabilize the newborn whilst the other professional inserts the naso-gastric feeding tube.
  Interventions: Other: Installation of a naso-gastric feeding tube
- Containing support with equipment (Other): Carried out by one healthcare Professional, who places the newborn in such a manner that he will be held in the optimum position (using a soft sheet) during the insertion of the naso-gastric feeding tube.
  Interventions: Other: Installation of a naso-gastric feeding tube

INTERVENTIONS:
Other: Installation of a naso-gastric feeding tube — Insertion of the feeding tube with skin-to-skin contact or whilst being held in the mother's arms, or by using the four hands technique or by performing positional support with appropriate equipment

SUMMARY:
Out of the most commonly performed procedures in neonates, naso-gastric tube insertion is rated as the fifth most painful. The pain is often under estimated due to the frequency with which the procedure is carried out. It has been shown that the environment in which the procedure is performed (e.g with skin to skin contact and specific positioning), reduces the discomfort felt by the newborn. However, this has not yet been proven with regards to naso-gastric tube insertion.

DETAILED DESCRIPTION:
Our clinical study (carried out in the Neonatology Unit of Mercy Regional Hospital) has shown that when positioning and other non drug related analgesic techniques are used, newborns undergoing naso-gastric tube insertion feel less pain.

Several different techniques were used, such as skin-to-skin contact with the mother and/or positioning the infant using appropriate equipment, or the "four hands" technique carried out by two health care professionals.

Neonatal unit staff were able to choose the method used depending on whether the mother was present at the time of the procedure.

In cases where the mother was absent, the "four hands technique" was favored, but in the presence of the mother skin-to-skin contact was preferable.

ELIGIBILITY:
Inclusion Criteria:

* Preterm baby born between the 32th and the 35th weeks of amenorrhea plus 6 days
* Prescription of enteral nutrition via naso-gastric tube
* Naso-gastric tube in-situ
* Informed consent of both parents

Exclusion Criteria:

For the newborn

* Under respiratory assistance
* With nasal or buccal malformation
* With abnormal heart rhythm or congenital heart disease
* With hemodynamic instability
* Transfer to type 3 neonatal unit
* With a DAN score > 0 before treatment
* With an umbilical venous catheter in-situ
* Fed with thickened milk
* Prescription of analgesic medications

For the parents

* Minor
* Under legal protection
* Difficulties which do not permit the mother to carry out skin-to skin contact or holding support

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

PRIMARY OUTCOMES:
Pain during insertion of the probe | Day 1
  Evaluation of the newborn's pain during insertion of the naso-gastric tube using the Premature Infant Pain Profile (PIPP) scale. The PIPP consists of 3 behavioral (facial actions: brow bulge, eye squeeze, and nasolabial furrow) and 2 physiological (heart rate and oxygen saturation) indicators, and 2 contextual [gestational age (GA) and behavioral state] variables that modify pain. In the same time, the heart rate and oxygen saturation of the newborns were measured using a pulse oximeter.

SECONDARY OUTCOMES:
Evaluation of pain using the DAN scale | Day 1
  This scale scores pain from 0 to 10, where 0 is no pain and 10 is maximum pain; it evaluates three items: facial expressions, limb movements and vocal expression.
Maternal satisfaction | Day 1
  Mother's satisfaction with regards to her involvement in the procedure. The questions are about her sense of usefulness during the probe, her knowledge of child's reaction and her desire to repeat the experience.
Professional's satisfaction | Day 1
  Health carers satisfaction during the procedure. The questions are about his appreciation of the effective management of the pain, the ease of installation, the benefits of the mother's presence and his desire to repeat the experience.
Duration of the Naso -gastric tube in situ | Day 7
  Lifetime of the probe after insertion
Procedure time | Day 1
  Time taken to insert the naso-gatric tube

CONTACTS AND LOCATIONS:
Locations (1):
- CHR Metz Thionville, Metz, France